CLINICAL TRIAL: NCT02162069
Title: Coronary and Structural Interventions - Transcatheter Aortic Valve Replacement
Acronym: CSI-TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Jochen Wohrle, Prof. Dr. Jochen Wöhrle, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSI TAVR 1.0
Record Dates: First submitted 2014-06-07; First posted 2014-06-12 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: TAVR
Oversight: Data Monitoring Committee: No

ARMS (1):
- transcatheter aortic valve replacement (Experimental): Patients receive transcatheter aortic valve replacement.
  Interventions: Device: CE certified transcatheter ( aortic valve replacement)

INTERVENTIONS:
Device: CE certified transcatheter ( aortic valve replacement) — Patients receive a transcatheter aortic valve replacement with CE certified transcatheter aortic valves.

SUMMARY:
To evaluate the long-term results after transcatheter aortic valve replacement

DETAILED DESCRIPTION:
Patients with transcatheter aortic valve replacement are followed for 5 years to demonstrate efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* aortic valve stenosis
* transcatheter aortic valve replacement

Exclusion Criteria:

* no written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2014-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Major adverse cerebral and cardiac events. | 1-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Wöhrle, MD, Principal Investigator — University of Ulm, Ulm, Germany
Locations (1):
- University of Ulm, Ulm, Germany

REFERENCES:
- [Background] Seeger J, Gonska B, Otto M, Rottbauer W, Wohrle J. Cerebral Embolic Protection During Transcatheter Aortic Valve Replacement Significantly Reduces Death and Stroke Compared With Unprotected Procedures. JACC Cardiovasc Interv. 2017 Nov 27;10(22):2297-2303. doi: 10.1016/j.jcin.2017.06.037. Epub 2017 Sep 13. PMID 28917515
- [Result] Seeger J, Kapadia SR, Kodali S, Linke A, Wohrle J, Haussig S, Makkar R, Mehran R, Rottbauer W, Leon M. Rate of peri-procedural stroke observed with cerebral embolic protection during transcatheter aortic valve replacement: a patient-level propensity-matched analysis. Eur Heart J. 2019 May 1;40(17):1334-1340. doi: 10.1093/eurheartj/ehy847. PMID 30590554
- [Derived] Vernikouskaya I, Bertsche D, Rottbauer W, Rasche V. Deep learning-based framework for motion-compensated image fusion in catheterization procedures. Comput Med Imaging Graph. 2022 Jun;98:102069. doi: 10.1016/j.compmedimag.2022.102069. Epub 2022 May 13. PMID 35576863
- [Derived] Seeger J, Gonska B, Rottbauer W, Wohrle J. New generation devices for transfemoral transcatheter aortic valve replacement are superior compared with last generation devices with respect to VARC-2 outcome. Cardiovasc Interv Ther. 2018 Jul;33(3):247-255. doi: 10.1007/s12928-017-0477-6. Epub 2017 Jun 22. PMID 28643214
- [Derived] Seeger J, Gonska B, Rottbauer W, Wohrle J. Outcome With the Repositionable and Retrievable Boston Scientific Lotus Valve Compared With the Balloon-Expandable Edwards Sapien 3 Valve in Patients Undergoing Transfemoral Aortic Valve Replacement. Circ Cardiovasc Interv. 2017 Jun;10(6):e004670. doi: 10.1161/CIRCINTERVENTIONS.116.004670. PMID 28566290
- [Derived] Seeger J, Gonska B, Rodewald C, Rottbauer W, Wohrle J. Impact of suture mediated femoral access site closure with the Prostar XL compared to the ProGlide system on outcome in transfemoral aortic valve implantation. Int J Cardiol. 2016 Nov 15;223:564-567. doi: 10.1016/j.ijcard.2016.08.193. Epub 2016 Aug 17. PMID 27561160
- [Derived] Wohrle J, Gonska B, Rodewald C, Seeger J, Scharnbeck D, Rottbauer W. Transfemoral Aortic Valve Implantation with the New Edwards Sapien 3 Valve for Treatment of Severe Aortic Stenosis-Impact of Valve Size in a Single Center Experience. PLoS One. 2016 Mar 22;11(3):e0151247. doi: 10.1371/journal.pone.0151247. eCollection 2016. PMID 27003573